CLINICAL TRIAL: NCT04678687
Title: Evaluation of Postmortem Biopsy Specimens of COVID-19 Cases
Brief Title: COVID-19 and Tissue Damage in Vital Organs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Mehmet Nuri Yakar, MD, PhD, Research Assistant, Dokuz Eylul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVID-19.PMB
Record Dates: First submitted 2020-12-02; First posted 2020-12-22 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Postmortem Changes
MeSH Terms: conditions — COVID-19; Postmortem Changes | interventions — Liver Extracts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 group (Other): Liver, lung, heart and kidney biopsies will be performed on each case in the COVID-19 group.
  Interventions: Procedure: Liver, lung, heart and kidney biopsy

INTERVENTIONS:
Procedure: Liver, lung, heart and kidney biopsy — Liver, lung, heart and kidney biopsies will be performed on each case in the COVID-19 group.

SUMMARY:
The study will be conducted in Dokuz Eylül University Hospital, COVID-19 (Coronavirus Disease 2019) intensive care unit. Three primary conditions will be sought for participants:

1. Cases whose treatment process resulted in death will be included in the study.
2. The cases must be confirmed with the diagnosis of COVID-19 by the RT-PCR (real time polymerase chain reaction) test.
3. The first-degree relatives must consent for the participation of the subjects in the study by their first-degree relatives.

In the study, samples will be taken from the liver, kidney, lung, and heart. The samples will be stored in a protective solution and sent to the pathology unit. The examinations will determine the microscopic damage to these organs caused by COVID-19.

Also, the presence of the SARS-CoV-2 (Severe Acute Respiratory Syndrome Coronavirus 2) will be investigated by RT-PCR in tissues. The presence of ACE-2 (angiotensin converting enzyme 2) receptor and SARS-CoV-2 nucleoprotein antibody will be investigated by histochemical examination in tissues.

DETAILED DESCRIPTION:
The cases whose treatment resulted in death at Dokuz Eylül University Research and Application Hospital Anesthesiology Intensive Care Unit and whose COVID-19 diagnosis was confirmed by the RT-PCR (real time polymerase chain reaction) test and gave written consent to the inclusion of the patient in the study by a first-degree relative will be included in the study. In the study, samples will be taken from 10 cases in total.

Age, gender, length of hospital stay, respiratory rate at the time of hospitalization, oxygene saturation on ICU admission and Horwitz ratio on ICU admission will be recorded. Also, the comorbidities of these cases, the interpretation of the computed tomography findings performed at the first admission to the hospital in terms of COVID-19, the RT-PCR results routinely sent for COVID-19 examination will be recorded in the case report form. Besides, all medical and supportive treatments applied during the intensive care treatment will be recorded. Liver and kidney function tests, inflammation and coagulation markers, hemoglobin level , and cardiac markers, which are routinely examined at the patient's admission to the intensive care unit, will be recorded.

Postmortem biopsy samples will be performed within 1 hour after the diagnosis of death is confirmed by the patient's doctor. The researchers will perform the procedures in the isolated room prepared for interventional procedures in intensive care. Researchers will wear personal protective equipment (cap, mask, goggles, gloves) before the procedure under the Ministry of Health's instructions.

Biopsy specimens will be taken from the lung, liver, heart, and kidney. Heart, liver, and kidney biopsies were performed as a core biopsy with tru-cut needles under ultrasonography guidance; lung biopsy will be performed by passing through the airway using biopsy forceps.

Each of the biopsy samples will be placed separately in 10 ml of 10% phosphate-buffered formalin solution. The containers will be disinfected with 80% alcohol. It will be placed in a closed zippered bag and kept at room temperature. It will be delivered to the pathology unit after 24 hours. The procedures as tissue cassette, extended tissue tracing, paraffin blocking, sectioning, and hematoxylin-eosin staining will be performed under biosafety level 2 rules in pathology. The cases will be coded as CVDPM-1... (Coronavirus Disease Postmortem 1...). Case report forms will be shared with researchers who will conduct pathological examination over the internet. Informed consent forms received from patients' relatives will be filed in the COVID-19 Intensive Care Unit.

Routine pathology sections will be evaluated in light microscopy according to the following criteria.

Lungs; alveolar epithelial cell damage, hyaline membrane formation, type 2 pneumocyte hyperplasia, diffuse alveolar damage, fibroblastic proliferation, fibrin accumulation, inflammatory infiltration, and the nature of inflammation Liver; lobular lymphocyte infiltration, centrilobular sinusoidal dilatation Kidney; diffuse proximal tubule damage, brushed edge loss, non-isometric vacuolar degeneration, necrosis, hemosiderin, pigmented cast, capillary plugs, vasculitis, intercalary inflammation, hemorrhage, Heart; acute ischemic injury, vascular pathology, inflammation Tissues will be tested for the presence of the SARS-CoV-2 virus by RT-PCR test. ACE2 receptor and SARS-CoV-2 nucleoprotein antibody will be examined by immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Cases 18 years and older than 18 years.
* Cases diagnosed with COVID-19 confirmed by PCR test.
* Cases whose treatment resulted in death.
* Cases that was allowed the participation in the study by signing the informed consent form by their first degree relatives.

Exclusion Criteria:

* Cases less than 18 years old.
* Cases for which the diagnosis of COVID-19 could not be confirmed.
* Cases for which informed consent could not be obtained.
* Cases whose treatment continues or results in healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
The level of histopathological changes | in three months after the participant's death
  In lung; alveolar epithelial cell damage, hyaline membrane formation, type 2 pneumocyte hyperplasia, diffuse alveolar damage, fibroblastic proliferation, fibrin accumulation, inflammatory infiltration and the nature of inflammation. In liver; lobular lymphocytic infiltration, centrilobular sinusoidal dilatation. In kidney; diffuse proximal tubule damage, brushed edge loss, non-isometric vacuolar degeneration, necrosis, hemosiderin, pigment cast, capillary plugs, vasculitis, interciliary inflammation, hemorrhage. In heart; acute ischemic injury, vascular pathology, inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Ali N Gökmen, MD, PhD, Principal Investigator — Dokuz Eylul University, Department of Anaesthesiology and Reanimation, Division of Intensive Care; Mehmet N Yakar, MD, PhD, Study Director — Dokuz Eylul University, Department of Anaesthesiology and Reanimation, Division of Intensive Care; Safiye Aktaş, MD, PhD, Study Director — Dokuz Eylul University, Oncology Institute, Department of Basic Oncology; Bilgin Cömert, MD, PhD, Study Director — Dokuz Eylul University, Department of Internal Medicine, Division of Intensive Care; Begüm Ergan, MD, PhD, Study Director — Dokuz Eylul University, Department of Chest Disease, Division of Intensive Care; Bişar Ergün, MD, PhD, Study Director — Dokuz Eylul University, Department of Internal Medicine, Division of Intensive Care; Fırat Bayraktar, MD, PhD, Study Chair — Dokuz Eylul University, Department of Internal Medicine, Division of Endocrinology and Metabolism; Eyüp S Uçan, MD, PhD, Study Chair — Dokuz Eylul University, Department of Chest Disease; Aylin Erol, Study Chair — Dokuz Eylul University, Oncology Institute; Özde E Gökbayrak, Study Chair — Dokuz Eylul University, Oncology Institute
Locations (1):
- Dokuz Eylul University, Izmir, Balçova, Turkey (Türkiye)